CLINICAL TRIAL: NCT00162708
Title: A Randomized Trial Evaluating a Very Intense Radiotherapy-Chemotherapy Regimen Versus a Very Accelerated Radiotherapy in Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Very Intense Radiotherapy-Chemotherapy Regimen in Advanced HNSCC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VADN3; GORTEC
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Oropharynx Cancer; Oral Cancer; Hypopharynx Cancer; Larynx Cancer
Keywords: Head and neck squamous cell carcinoma; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Fluorouracil

INTERVENTIONS:
Procedure: Radiotherapy 62-64 Gy in 5 W (31-32 f. of 2 Gy BID)
Procedure: Radiotherapy 62-64 Gy in 22-23 D (31-32 f of 2 Gy BID)
Drug: CDDP, 5 Fu

SUMMARY:
Altered fractionated radiotherapy and concomitant radio-chemotherapy have been shown to be two possibilities for improving efficacy of radiotherapy in locally advanced head and neck carcinomas. In this multicentric study, we tested the hypothesis that accelerated radiotherapy could be delivered concomitantly with conventional high doses of CDDP-5FU, aiming to improve both local control and on distant metastases as compared to very accelerated radiotherapy.

DETAILED DESCRIPTION:
Patients with a palpable N2b-c or N3 HNSCC strictly unresectable were randomized to receive either accelerated RT-CT delivering to the primary tumor 62-64 Gy / 5 weeks in 31-32 fractions of 2 Gy BID or very accelerated RT delivering 62-64 Gy in 31-32 fractions of 2 Gy BID and 22-23 days. In the accelerated RT-CT arm, 3 cycles of CDDP 100 mg/m2 were delivered at day 1, 16, 32 and 2 cycles of 5 Fu 1000 mg/m2 day 1 to 5 and 31 to 35. One month after completion of the concomitant RT-CT, 2 additional cycles of CDDP-5FU were given in patients responding (> 50%) to the initial course of RT-CT. The end points were event free survival and survival.

ELIGIBILITY:
Inclusion Criteria:

* palpable N2b-c or N3 (UICC 1997) squamous cell carcinoma of the head and neck (oropharynx, oral cavity, hypopharynx or larynx)
* primary tumor and / or nodal extension strictly inoperable due to the extension of the disease
* performance status of 0 to 2 (WHO scoring system)
* renal/liver/cardiac functions and blood counts compatible with the use of CDDP and 5-FU
* signed inform consent

Exclusion Criteria:

* distant metastasis
* previous history of cancer
* previous radiotherapy or chemotherapy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1996-07

PRIMARY OUTCOMES:
Event free survival (event = progressive disease or relapse or or death from any cause)

SECONDARY OUTCOMES:
Survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourhis, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Michel Lapeyre, Principal Investigator — Centre Alexis Vautrin; Jacques Tortochaux, Principal Investigator — Centre Jean Perrin
Locations (3):
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Alexis Vautrin, Nancy
  - Institut Gustave Roussy, Villejuif